CLINICAL TRIAL: NCT03062488
Title: Emergence Agitation and Pain Scores in Pediatric Patients Following Sevoflurane Anesthesia When Comparing Single-modal Versus Multi-modal Analgesia for Routine Ear-nose-throat (ENT) Surgery, a Multi-center Double-blinded Study
Brief Title: Emergence Agitation and Pain Scores in Pediatrics When Comparing Single-modal vs Multi-modal Analgesia for ENT Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB1074554
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2017-08

CONDITIONS: Emergence Agitation; Pain
MeSH Terms: conditions — Emergence Delirium; Pain | interventions — Acetaminophen; Fentanyl

STUDY DESIGN:
Intervention Model Description: Study Design:
  1. Prospective Randomized Study
  2. Study Period: August 2017 - December 2017
  3. Potential participants: 375 - 475 based on 20-25% of 4,459 ENT patients in 2016
  4. Study Population: 50 pediatric patients in each group between 24 months through 7 years of age undergoing adenoidectomy or tonsillectomy with or without adenoidectomy Total Number of Patients: 150
Who Masked: Participant, Care Provider, Investigator
Masking Description: all patients will receive a de-identified PO syrup. The syrup will be prepared by the pharmacy and will contain acetaminophen (15 mg/kg) for the PO acetaminophen group and placebo flavored syrup for the other two groups. This approach will maintain blindness of the peri-operative staff, and patients/parents., all children will receive fentanyl 2 mcg/Kg IV. Intra-op anesthesia team will be blinded to the use of non-opioid IV analgesia and will administer a pharmacy prepared de-identified infusion following intubation that will consist of saline placebo for control groups and IV acetaminophen (15 mg/kg) for the IV acetaminophen group. ,
  :A blinded PACU nurse will record degree of agitation using the PAED scale on admission to the PACU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- opioid only (Active Comparator): 2 mcg/Kg of fentanyl
  Interventions: Drug: Fentanyl
- opioid plus PO analgesic (Active Comparator): 2 mcg/Kg of fentanyl plus PO acetaminophen 15 mg/Kg
  Interventions: Drug: Fentanyl; Drug: PO acetaminophen
- opioid plus IV acetaminophen (Active Comparator): 2 mcg/Kg of fentanyl plus 15mg/Kg of IV acetaminophen
  Interventions: Drug: IV acetaminophen; Drug: Fentanyl

INTERVENTIONS:
Drug: IV acetaminophen — multi-modal analgesia with IV acetaminophen
  Other Names: Ofirmev
  Arms: opioid plus IV acetaminophen
Drug: Fentanyl — single modal analgesia
  Other Names: duragesic
Drug: PO acetaminophen — multi-modal analgesia with PO acetaminophen
  Other Names: tylenol
  Arms: opioid plus PO analgesic

SUMMARY:
The purpose of this study is to compare the incidence of EA in pediatric patients undergoing minor ENT surgery under Sevoflurane and compare opioid-only based intra-operative analgesia to multi-modal analgesia consisting of opioid and IV acetaminophen or PO acetaminophen regimen using a validated and standardized EA measurement tool, the Pediatric Anesthesia Emergence Delirium (PAED) scale. The post operative pain scores will be measured in all patients by post-op recovery staff using FLACC Score/Wong-Baker FACES (patients 24 months up to 7 years of age) or Numeric Pain Score for patients 7 years of age. The pre-operative, surgery, anesthesia and post-operative staff will be all blinded.

DETAILED DESCRIPTION:
Place of Study:

Nemours Children's Hospital, Orlando, Florida (Primary Site) Wolfson Children's Hospital, Jacksonville, Florida (Nemours Jacksonville Satellite Site)

Study Design:

Prospective Randomized Study Total Number of Patients: 150

Methods and Materials: 150 patients will be randomly divided into three groups of 50 patients. Each group will receive sevoflurane induction and maintenance of anesthesia. Sevoflurane, currently the most commonly used agent for inhalational induction, will be used for induction of anesthesia, as it is less irritating to the tracheobronchial tree than other volatile anesthetic agents and is considered the standard for pediatric induction anesthesia. These three groups, (study arms), are identified as follows:

Group A: multi-modal analgesia of IV fentanyl plus IV acetaminophen and oral placebo Group B: multi-modal analgesia of IV fentanyl plus PO acetaminophen and IV placebo Group C: single modal analgesia of IV fentanyl plus oral placebo and IV placebo Pre-operative procedures: The Research Pharmacy will have the following standards for randomization: prior to patient surgery date; the pharmacy will assemble study kits to contain the appropriate drug products based on the 3 randomization scenarios: A. IV Tylenol and Oral Placebo, B. IV Placebo and Oral Tylenol, or C. IV Placebo and Oral Placebo. The kits will be kept in the pharmacy and identified in a blinded fashion from other study team members. On the day of surgery, (patient dosing day), blinded study team member will provide the signed study consent to pharmacist, along with the patient's weight to be used in calculating dosages of study drug. The pharmacist will then assign the patient to 1 of 3 study arms, in a random approach. Randomization will be performed by using a method based on the biased coin method using a dynamic urn technique. Once the study arm has been determined, the corresponding kit will be used to prepare the study drugs by patient weight. The blinded, randomized study kit information will be kept in a locked Excel spreadsheet, with password access, only available to pharmacy team members. All study drugs will be checked and verified by a licensed pharmacist prior to dispensing to a blinded study team member.

None of the study patients will receive premedication for sedation. Premedication is not a standard treatment at Nemours Children's Hospital (NCH) as NCH allows parental presence during induction of anesthesia to facilitate the transport of the patient to the operating room and decrease separation anxiety. Wolfson Children's Hospital will allow parental presence for study patients. Parental presence is an appropriate substitute for sedation premedication. In the pre-operative area, all patients will receive a de-identified PO syrup. The syrup will be prepared by the pharmacy and will contain acetaminophen (15 mg/kg -160mg/5mL Manufacturer: Major Pharmaceuticals), for the PO acetaminophen group and placebo flavored syrup (Manufacturer: Humco, Ingredients: Sucrose 82.3%, Purified Water, Artificial Flavors, 0.1% Sodium Benzoate as a preservative, Critic Acid, FDC Red #40, and inert ingredients), for the other two groups. This approach will maintain blindness of the peri-operative staff, and patients/parents/guardians.

Intraoperative Procedures and Administration of intra-op analgesia: Before induction of anesthesia the pre-induction vital signs will be reviewed and ASA standard monitors will be applied. Standard ASA monitors include blood pressure, ECG, pulse oxymetry, etCO2

Measurement, respiratory rate and temperature. Induction of anesthesia will be accomplished via inhalation of sevoflurane (8 vol%) in nitrous oxide (70%) and oxygen (30%) at a fresh gas flow of 10 Lpm. An IV will be established and propofol 2mg/Kg will be administered to facilitate endotracheal intubation. After intubation, all children will receive fentanyl (West- Ward Pharmaceuticals) 2 mcg/kg. IV Fentanyl is considered standard of care for analgesia regimen for these types of surgery. Intra-op anesthesia team will be blinded to the use of non- opioid IV analgesia and will administer a pharmacy prepared de-identified infusion (pharmacy will blind the IV formulation of acetaminophen and all pharmacy formulations will follow regulation 797 compounding standards), following intubation that will consist of 0.9% normal saline (Baxter Pharmaceuticals), placebo for control groups and IV acetaminophen (15 mg/kg, - 1000mg/100 cc Mallinckrodt Pharmaceuticals) for the IV acetaminophen group. The maximum single dose will be 750 mg with a 24-hour maximum dose not to exceed 3,750 mg in this 24-hour period. The product will infuse for 15 minutes as recommended by the manufacturer. For maintenance of anesthesia, children will receive sevoflurane (maximum of 2.0±0.2 MAC, age adjusted) with a constant fresh gas flow of 2 L/min (maximum FIO2 of 30% air mixed with oxygen), using a semi-closed circle breathing system. Ventilation will be controlled to maintain normocapnia (ET-CO2 32-38 mmHg). Additional doses of fentanyl can be administered, per anesthesiologist's discretion, in all groups by increments of 0.5 mcg/Kg IV per dose for hemodynamic response to surgical stimulation greater than 20% above baseline. Removal of the mouth gag for tonsillectomy/tonsillectomy and adenoidectomy/adenoidectomy will be defined as the end of surgery. At this point, inhalation anesthetic will be discontinued. Fresh gas flow will be increased to 8 Lpm, 100% oxygen. Tracheal extubation will be performed when normal ventilation is achieved and cough or gag reflex is regained.

Screening/Consent Process: Potential participants will be identified and receive basic information about the study and enrollment criteria at ENT clinic by participating ENT surgeons. A copy of an unsigned consent will be given to the families who are interested in participating in the study. Anesthesiologists, will obtain PP consent and Assent for eligible children. A signed and dated copy of all consents forms will be given to the parents.

Intraoperative Standardization and Procedures: The surgical technique will be standardized and a limited group of two surgeons per clinical site that share same surgical technique which will be agreed upon at the start of the clinical phase. This technique will consist of only Teflon blade cautery and will require no peri-tonsilar local anesthetic injection. The number of anesthesia providers involved in the study will be limited to two anesthesiologists per clinical site.

The post-operative pain management approach will be restricted to fentanyl (0.5 mcg/Kg IV/dose titrated to effect) for moderate to severe pain. Ibuprofen (10mg/Kg) PO will be ordered for mild to moderate post- op pain. Post-op recovery staff will be limited to a maximum of three trained PACU nurses per site and will use FLACC Scale for age 24 month to 4 years of age and sedated patients at time of assessment, Wong-Baker FACES for patients 4 to 7 years of age and non-verbal patients and Numeric Pain Score for patients equal/greater than 7 years of age to assess level of pain. Episodes of clinical emergence agitation/delirium (EA), will receive rescue treatment. This treatment will consist of 0.5 - 1.0 mcg/Kg IV dexmedetomidine.

Age, gender, height, weight, procedure, duration of surgery, intra-op agents used, exposure and time of discontinuation of anesthesia to extubation will be documented for each patient. A blinded PACU nurse will monitor the patient. The Post-anesthesia unit monitoring standards consist of ECG, Blood Pressure, pulse-oxymetry and respiratory rate every 5 minutes times 3 and every 15 minutes thereafter until discharge. Temperature will be obtained upon arrival to unit and every hour or as needed. All patients will be evaluated for the Aldrete Score which assesses readiness for discharge from post-anesthesia care unit. The PACU nurse will record degree of agitation using the PAED scale and measure and record the pain scores using either the FLACC for patients 24 months to 4 years of age and patients who are sedated at time of assessment, Wonk-Baker FACES for patients 4 to 7 years of age and non-verbal patients and Numeric Pain Scores for patients equal/greater than 7 years of age upon admission to the PACU and every 15 minutes for approximately 1 hour after admission, or until discharge from the PACU, whichever comes first. These nurses will all be experienced in the use of PAED scale. There will be three; two-hour study training sessions at each clinical site for PACU participating nurses. PACU nurses assigned to this study will be selecting the Modified Aldrete scores (respiration, O2saturation, consciousness, circulation, activity) and documenting adverse events

Monitoring Procedures:

The investigative team assures that informed consent is obtained prior to performing any research procedures, that all subjects meet eligibility criteria, and that the study is conducted according to the IRB-approved research protocol.

Collection and Reporting of SAEs and AEs:

For this study, the following standard AE definitions are used:

Adverse event: Any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.

Serious Adverse Event: Any AE that results in any of the following outcomes:

* Life-threatening event
* Event requiring inpatient hospitalization or prolongation of hospitalization
* Death
* Congenital anomaly
* Persistent or significant disability/incapacity
* Required intervention to prevent permanent impairment/damage

AEs identified will be captured in real time as they become known. AEs that result in visits to the ED and/or outpatient clinics will be monitored at each site through their readmission- monitoring program and reported to the department of Anesthesiology by the quality and safety officer. In addition, all AEs are reported in Orlando according to the Nemours IRB AE reporting guidelines and in Jacksonville, according to the Baptist Health IRB AE guidelines.

Treatment of AEs:

In case of a symptomatic event where a severe adverse event or any SAE is noticed, the blinding can be broken by accessing a sealed envelope that contains the assigned drugs in the randomization process and appropriate treatment will be instituted. These patients will be withdrawn from the study but the clinical and research team will continue to collect safety information. This data will be included in the safety database and reported during monthly meetings. Nemours will assure that the participant receives treatment, if needed , for study- related injuries.

Ameliorating Measures:

Episodes of clinical emergence agitation/delirium (EA), will receive rescue treatment. This treatment will consist of 0.5 - 1.0 mcg/Kg IV dexmedetomidine as previously stated.

All patients will be instructed not to start the next dose of acetaminophen until 6 hours after last administered dose. This dose correlates to the time of intra-operative IV infusion administration.

All discharged patients will receive a call within 24 hours of surgery for follow-up.

* Compliance of regulatory documents as well as study data accuracy and completeness, will be monitored through an internal study team quality assurance process.
* Confidentiality throughout the trial is maintained by securing identifiable participant data in secured,

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 24 months through 7 years of age
2. Patients who weigh <50 kg
3. Patients who are able to take PO medications
4. Patients who are ASA Classification I and II
5. Patients who are found to be a candidate after clinical review of detailed History and Physical Exam, review of Polysomnogram or Pediatric Sleep Questionnaire
6. Patients who are scheduled for routine adenoidectomy or tonsillectomy with or without adenoidectomy not in conjunction with another invasive or diagnostic procedure
7. Patients who meet clinical indications for surgery
8. Family and patient must be proficient in English to understand consent, post-operative instructions, and facilitate the assessment after emergence of anesthesia

Exclusion Criteria:

1. Children with a history of developmental delay or psychological disorders that may be at higher risk for EA as determined by study physician after review of history and problem list in EMR
2. Patients with previous hypersensitivity to oral or intravenous acetaminophen, fentanyl or any of its components or ingredients in placebo,
3. Patients with severe hepatic impairment or severe active hepatic disease
4. Patients with previous history of Malignant Hyperthermia or susceptibility to volatile anesthetics agents like sevoflurane
5. Any patient who weighs >50 Kg.
6. Any patient that requires premedication. Versed may contribute to an increase in EA. Premedication is reserved when parental presence is not feasible or for very anxious children.
7. Patients unable to take PO (acetaminophen or placebo) will be excluded from the study.
8. Children with severe symptomatic sleep apnea that require post-operative hospitalization.
9. Severe symptomatic sleep apnea is defined as a- patients who has a pre-operative polysomnogram and a calculated Apnea-Hypoxia Index greater than 10 b- patients with high scoring in Pediatric Sleep Questionnaire (PSQ)
10. Patients with severe symptoms and findings in physical exam that require post-operative hospital admission.
11. Patients and/or families not proficient in English
12. Participant is currently participating or has within the previous 30 days, participated in another clinical trial/research study

Ages: 24 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Archilla, MD, Principal Investigator — Nemours Children's Hospital
Locations (1):
- Nemours Children's Specialty Care, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Place of Study: Nemours Children's Hospital, Orlando, FL and Wolfson Children's Hospital, Jacksonville, FL
  Design:
  Prospective Randomized Study Study Period: October 2017-March 2018 Population: 50 pediatric patients in each group between 24 months through 7 years of age undergoing adenoidectomy or tonsillectomy with or without adenoidectomy
Pre-assignment Details: No events. Patients were screened prior to pre-enrollment.
Period: Overall Study
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen
Started | 51 | 51 | 41
Completed | 51 | 51 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen | Total
Number analyzed (Participants) | 51 | 51 | 41 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.49 (1.5) | 4.9 (1.58) | 4.61 (1.28) | 4.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 19 | 74
  Male | 22 | 25 | 22 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 12 | 42
  Not Hispanic or Latino | 37 | 35 | 29 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kg] — Measured in Kilograms of weight
  Kg | 19.99 (5.81) | 21.79 (5.94) | 20.94 (5.39) | 20.9 (5.7)
body mass index [Mean (Standard Deviation); unit: Kg/m²] — a weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters and used as an indicator of obesity and underweight.
  Kg/m² | 16.59 (2.31) | 17.21 (3.35) | 16.70 (2.67) | 16.8 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Emergence Agitation (EA) as Measured by Standardized PAED Scale
Description: Post Anesthesia Emergence Delirium (PAED) Scale 0 - 20. EA defined as a score equal or greater than 12
Time Frame: first 60 minutes of recovery post anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen
Number analyzed (Participants) | 51 | 51 | 41
score on a scale | 5.3 (2.77) | 4.99 (2.6) | 6.29 (2.85)

2. Secondary Outcome: Post Operative Pain
Description: Measured on scale of 0-10 0-3 = mild pain 4-6 = moderate pain 7-10 = severe pain Tools used for each age subgroup: FLACC Score for patients 24 months to 4 years of age and sedated patients at time of assessment, Wong-Baker FACES for patients between 4 and 7 years of age, and Numeric Pain Scores for patients equal/greater than 7 years of age
Time Frame: Average in first 60 minutes of recovery post anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen
Number analyzed (Participants) | 51 | 51 | 41
score on a scale | 2.58 (1.86) | 2.56 (1.60) | 2.51 (1.83)

3. Secondary Outcome: Post Operative Fentanyl Consumption
Description: Post operative administration of fentanyl in micrograms per Kilogram of weight after intra-operative pain management in the Post Anesthesia Care Unit (PACU)
Time Frame: first 60 minutes in the PACU
Measure: Mean (Standard Deviation); unit: microgram per Kg of weight
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen
Number analyzed (Participants) | 51 | 51 | 41
microgram per Kg of weight | 0.64 (0.50) | 0.72 (0.61) | 0.58 (0.52)

ADVERSE EVENTS:
Time Frame: 24 hours. Any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure observed or measured from administration of pre-operative medication, intra-operative and immediate [postoperative periods until 24 to 48 hour follow up phone call
Arm/Group | Opioid Only | Opioid Plus PO Analgesic | Opioid Plus IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/41
Other Adverse Events (participants affected / at risk) | 13/51 | 17/51 | 15/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Only (N=51) | Opioid Plus PO Analgesic (N=51) | Opioid Plus IV Acetaminophen (N=41)
Shivering (General disorders) | 0 (0) | 1 (1) | 0 (0)
Breath Holding (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Excessive Secretions (General disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Emergence Agitation (EA) Pharmacological Treatment (Psychiatric disorders) | 3 (3) | 5 (5) | 8 (8) — Patients who received pharmacological treatment for this
Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Oral Intake (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Excessive (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03062488/Prot_SAP_002.pdf
  • Informed Consent Form (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03062488/ICF_003.pdf